CLINICAL TRIAL: NCT02017314
Title: Correlation of Postoperative VAS Values and Body Mass Index in Patients Undergoing Abdominal Surgery: A Clinical Trial
Brief Title: VAS Correlation With BMI
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Guniz M.Koksal, Assc.Prof, Istanbul University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 830458909
Record Dates: First submitted 2013-12-08; First posted 2013-12-20 (Estimated); Last update posted 2013-12-20 (Estimated); Status verified 2013-12

CONDITIONS: Morbid Obesity
Keywords: morbid obesity; postoperative pain
MeSH Terms: conditions — Obesity, Morbid; Pain, Postoperative | interventions — Morphine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Group 5 (Active Comparator): Patients with BMI > 50
  Interventions: Drug: Morphine
- Group IV (Active Comparator): Patients with BMI between 40 and 49.9
  Interventions: Drug: Morphine
- Group III (Active Comparator): Patients with BMI between 35 and 39.9
  Interventions: Drug: Morphine
- Group II (Active Comparator): patients with BMI between 30 and 34.9
  Interventions: Drug: Morphine
- Group I (Active Comparator): Patients with BMI <30
  Interventions: Drug: Morphine

INTERVENTIONS:
Drug: Morphine

SUMMARY:
The aim of the study is to observe if any correlation between Body mass index and VAS values exists in patients who has gone under abdominal surgery.

Group I : Patients with BMI<30 Group II: Patients with BMI between 30 and 34.9 Group III: Patients with BMI between 35 and 39.9 Group IV: Patients with BMI between 40 and 49.9 Group V : Patients with BMI >50

After the end of surgery patients will be extubated and in the recovery room morphine PCA (patient-controlled analgesia) treatment will be started according to their adjusted body weight. When VAS values over 4,10 mg/kg Paracetamol IV will be used as an escape treatment. VAS values and Delivery and Demand of the PCA and additional need for analgesics will be recorded in the first 48 hours.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing abdominal surgery and who will be given PCA treatment for postoperative pain.

Exclusion Criteria:

* patients younger than 18 years old, patients with uncompensated diabetes or related polyneuropathy, patients receiving antidepressants or have a diagnosis of depression

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2013-11; Primary Completion 2014-03 (Estimated); Study Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
Pain Scores on the Visual Analog Scale | 48 hours
  Correlation between the VAS Scores and BMI will evaluated

CONTACTS AND LOCATIONS:
Locations (1):
- Cerrahpasa Medical School, Istanbul, Marmara, Turkey (Türkiye)

REFERENCES:
- [Background] Choi YK, Brolin RE, Wagner BK, Chou S, Etesham S, Pollak P. Efficacy and safety of patient-controlled analgesia for morbidly obese patients following gastric bypass surgery. Obes Surg. 2000 Apr;10(2):154-9. doi: 10.1381/096089200321668703. PMID 10782177